CLINICAL TRIAL: NCT03531047
Title: A Prospective, Controlled Study of Refractive Corneal Cross-linking for Progressive Keratoconus
Brief Title: Refractive Corneal Cross-linking for Progressive Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORD1003
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Keratoconus
Keywords: progressive; cross-linking; customised; refractive
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractive CXL (Experimental): Tomography-customised CXL
  Interventions: Procedure: Customised CXL

INTERVENTIONS:
Procedure: Customised CXL — As for standard CXL, following mechanical removal of the corneal surface layer (epithelium), 0.1% riboflavin drops will be applied every 2 minutes for 10 minutes prior to ultraviolet A (UVA) irradiation - UVA power, distribution and timing as determined by analysis of Pentacam tomography scans. A bandage contact lens will be applied to encourage regrowth of the corneal surface and reduce post-operative pain.
  Other Names: Riboflavin drops (drug): Vibex Rapid (Avedro Inc.)

SUMMARY:
Young patients with keratoconus face two problems: disease progression and corneal shape irregularity. Both underlie the 20% rate of corneal transplantation in keratoconics required to maintain useful vision.

Corneal collagen cross-linking (CXL) is a now the gold-standard treatment to halt disease progression. The aim is to strengthen the cornea to prevent further shape deterioration. For patients whose quality of vision has already suffered, standard CXL can generally only prevent further deterioration, rather than improving vision. Refractive CXL, a new iteration of CXL in which a bespoke treatment pattern is applied to the cornea, aims to smooth out surface irregularities thereby improving vision.

This primary objective of this study is to compare the visual outcome in patients with progressive keratoconus treated with refractive CXL, as compared with historical controls treated with standard CXL.

DETAILED DESCRIPTION:
Irregular astigmatism (irregular corneal shape leading to irregular focus) is a common cause of failure to achieve an adequate spectacle correction for many patients with corneal disease. For patients affected, rigid gas permeable contact lenses are the only means of visual rehabilitation. Not all patients tolerate rigid contact lens wear, and those that do are often uncomfortable and have a restricted wearing time.

Keratoconus, in which the corneal shape becomes progressively steeper and more irregular in the 2nd to 4th decades of life, is a common cause of irregular astigmatism. Disease progression in keratoconus can be stabilised with corneal collagen cross-linking (CXL), effective in 90% of cases. Pre-existing irregular astigmatism often remains after CXL, with many patients requiring rigid gas permeable contact lenses to regain good vision.

The investigators have recently demonstrated improvements in vision following simultaneous combined cross-linking with laser refractive surgery (TransPRK/CXL). The excimer laser is used to create a smoother, more regular focusing shape on the cornea to improve the quality of vision achieved in spectacles. Although effective, the downsides of using this approach are both the cost and limited availability of excimer laser equipment in the National Health Service (NHS) in the United Kingdom. Also, excimer laser smoothing works by removing corneal tissue. It is not yet known whether this tissue removal will have any detrimental effect on corneal shape stability post CXL.

As a cheaper and potentially more widely accessible alternative, refractive CXL aims to regularise the corneal surface by applying a bespoke treatment pattern based on pre-operative corneal surface shape (topography) scans. At least two-thirds of patients undergoing standard CXL already have impaired vision at the time treatment. The investigators are aiming to offer these patients both long-term stability of their keratoconus and an improvement in vision in a single treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with progressive stage I - III keratoconus
* Corrected distance visual acuity (CDVA) < 0.00 logMAR

Exclusion Criteria:

* Patients under the age of 18 years
* Active ocular surface disease
* Minimum corneal thickness < 375 µm
* Vulnerable groups
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Change in corrected distance visual acuity | 24 months
  LogMAR corrected vision in spectacles

SECONDARY OUTCOMES:
Change in uncorrected distance visual acuity | 24 months
  LogMAR uncorrected vision without spectacles
Manifest refraction | 24 months
  Spectacle prescription
Tomography | 24 months
  Corneal Pentacam indices
Rates of keratitis | 24 months
  Complications of CXL

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Gore, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gore DM, Shortt AJ, Allan BD. New clinical pathways for keratoconus. Eye (Lond). 2013 Mar;27(3):329-39. doi: 10.1038/eye.2012.257. Epub 2012 Dec 21. PMID 23258309
- [Result] O'Brart DP, Chan E, Samaras K, Patel P, Shah SP. A randomised, prospective study to investigate the efficacy of riboflavin/ultraviolet A (370 nm) corneal collagen cross-linkage to halt the progression of keratoconus. Br J Ophthalmol. 2011 Nov;95(11):1519-24. doi: 10.1136/bjo.2010.196493. Epub 2011 Feb 24. PMID 21349938